CLINICAL TRIAL: NCT01226563
Title: A Placebo Controlled, Multicenter, Randomized Double Blind Trial to Evaluate the Safety and Effectiveness of IK-5001 for the Prevention of Remodeling of the Ventricle and Congestive Heart Failure After Acute Myocardial Infarction
Brief Title: IK-5001 for the Prevention of Remodeling of the Ventricle and Congestive Heart Failure After Acute Myocardial Infarction
Acronym: PRESERVATION-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bellerophon BCM LLC (Industry)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IK-5001-VENREM-201
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2018-07

CONDITIONS: Acute Myocardial Infarction; Congestive Heart Failure; ST-Elevation Myocardial Infarction
Keywords: STEMI; Acute Myocardial Infarction; Congestive Heart Failure; Left Ventricular Remodeling; Devices, Medical
MeSH Terms: conditions — Heart Failure; ST Elevation Myocardial Infarction; Ventricular Remodeling | interventions — Abortion, Induced

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-controlled trial to evaluate the effects of IK-5001. 306 trials randomized 2:1 active vs placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: randomized 2:1 active vs placebo
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IK-5001 (Experimental): IK-5001 Sodium Alginate Calcium Gluconate intracoronary injection
  Interventions: Device: IK-5001
- Saline Solution (Placebo Comparator): Saline Solution intracoronary injection
  Interventions: Device: Saline Solution

INTERVENTIONS:
Device: IK-5001 — 4 mL (+/- 0.2 mL) administered through intracoronary slow bolus injection over 15 to 30 seconds at least 2 days after PCI but within 5 days of onset of symptoms.
  Other Names: Sodium Alginate Calcium Gluconate; BIOABSORBABLE CARDIAC MATRIX (BCM)
  Arms: IK-5001
Device: Saline Solution — 4 mL (+/- 0.2 mL) slow bolus, intracoronary injection of saline solution will be administered over 15 to 30 seconds at least 2 days after percutaneous coronary intervention (PCI) but within 5 days of onset of symptoms.
  Arms: Saline Solution

SUMMARY:
The primary objective is to evaluate the safety and effectiveness of the IK-5001 device for the prevention of ventricular remodeling and congestive heart failure when administered to subjects who had successful percutaneous coronary intervention with stent placement after ST segment elevation MI (STEMI).

DETAILED DESCRIPTION:
Heart failure is a significant problem, and carries substantial mortality. According to studies, left ventricular (LV) remodeling contributes independently to heart failure progression. Prevention and reversal of LV remodeling are correlated with decreased risk of death and heart failure events. IK-5001 is an implantable device to be used in subjects with recent myocardial infarction (MI). The IK-5001 device has been shown to directly halt the remodeling process that occurs following acute MI. IK-5001 replaces the damaged extracellular matrix (ECM) that has degraded during infarction, supports the damaged myocardial tissue, prevents local dyskinesis, and decreases wall stress. Because of its minimal interaction with the myocardium, its mechanism of action, its lack of specific pharmacologic activity and its elimination behavior, IK-5001 is a medical device in concurrence with the Global Harmonization Task Force's harmonized definition for medical devices.

ELIGIBILITY:
Inclusion criteria:

Subjects must meet all of the following inclusion criteria to participate in this trial:

1. The subject is ≥ 18 years of age.
2. The subject has given informed consent.
3. The subject has experienced a large STEMI defined by the following criteria:

   Peak cardiac enzyme value within 48 hours of symptom onset as follows:
   * Creatine kinase MB fraction (CK-MB) > 30 x the upper limit of normal OR
   * Troponin I > 200 x upper limit of normal OR
   * Troponin T > 60 x the upper limit of normal

   AND at least 1 of the following 3 criteria:
   * Delayed presentation with PCI > 6 hours from onset of symptoms
   * Significant new Q waves in ≥ 2 anterior leads or anterior ST segment elevation of at least 3 mm persistent at 24 hours after PCI
   * New onset of CHF (Killip class 3-4) or cardiogenic shock persistent at 24 hours after PCI

   AND at least 1 of the following 2 criteria:
   * MI ≥ 20% by Single Photon Emission Computed Tomography scan (SPECT) or cardiac Magnetic Resonance Imaging (MRI) with defect in the appropriate distribution
   * Ejection fraction ≤ 35% with wall motion abnormality in the appropriate distribution at baseline imaging assessment
4. The subject has had successful PCI with stent within 48 hours of symptom onset, and residual stenosis less than 20% in the infarct related artery and greater than or equal to thrombolysis in myocardial infarction (TIMI) 2 flow. Subjects undergoing rescue PCI after thrombolysis or delayed presentation with ongoing ischemia may be enrolled.
5. For Germany only: Patients determined to have Killip class 4 at time of device deployment are not eligible for randomization.
6. For Germany only: If SPECT is used for determination of MI size in order to meet inclusion criteria, the SPECT must have been previously performed as part of standard clinical care. SPECT is not to be performed solely to qualify a patient for this study in Germany.

Exclusion criteria:

Subjects will be excluded from participating in this trial if ANY of the following exclusion criteria are met:

1. Any subject with cardiogenic shock requiring mechanical ventilation or mechanical support at the time of deployment. Subject must be off mechanical support prior to deployment.
2. Need for urgent coronary artery bypass graft (CABG)
3. Clinically significant valvular heart disease with planned surgical correction or transcatheter aortic valve implantation (TAVI)
4. Uncontrolled ventricular arrhythmias
5. Renal insufficiency with a calculated creatinine clearance of less than 30 mL/ minute. See Appendix A for determining estimated creatinine clearance.
6. Clinically significant hepatic insufficiency
7. Inadequate imaging windows (defined as the inability to visualize the endocardial border of at least 16 of the 17 segments in both the apical four chambers and apical two chamber views without foreshortening) or arrhythmia that would preclude adequate 3D imaging on transthoracic echocardiography at the local baseline echo assessment
8. Non-ambulatory prior to the index MI
9. The subject has participated in another trial of an investigational agent within 30 days prior to randomization.
10. Subject has received resorbable stent as part of PCI.
11. The subject is pregnant or breastfeeding. Women of child-bearing potential will have a negative urine pregnancy test prior to randomization.
12. Any other concurrent condition that, in the opinion of the investigator, would prevent completion of the clinical trial, including inability to comply with follow up requirements.
13. For Germany only: In the investigator's opinion, the patient is not expected to survive ≥12 months.
14. For Germany only: 24 hours prior to device deployment, the patient has a serum calcium level greater than the upper limit of normal as determined by the local laboratory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2012-04; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Left Ventricular End Diastolic Volume Index | Baseline, 6 Months
  Anatomic measurement of left ventricular end diastolic volume index (LVEDVI) assessed through echocardiogram.

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionaire | Baseline (prior to index STEMI), 1, 3, 6 and 12 month follow-up visits
  Patient reported outcomes (PROs) using The Kansas City Cardiomyopathy Questionaire (KCCQ) score - a validated disease-specific self-administered 23-item questionnaire that will be used to quantify symptoms, function, and quality of life of subjects.
Six minute walk test | Baseline (prior to discharge STEMI), 1, 3, 6 and 12 month follow-up visits
  The six minute walk test (6MWT) is used for measuring the response to medical interventions in subjects with moderate to severe heart disease, functional status of subjects, as well as a predictor of morbidity and mortality
New York Heart Association (NYHA) functional classification (Physician reported) | Baseline (prior to index STEMI), 1, 3, 6 and 12 month follow-up visits
  New York Heart Association (NYHA) classification assessed by physician will be categorized by Class (Class I - IV)
Cardiovascular death, non-fatal heart failure events or cardiovascular hospitalizations | 5 Years
  Time to cardiovascular death, non-fatal heart failure events or cardiovascular hospitalizations adjudicated by a Clinical Events Committee
Re-hospitalization due to any cardiovascular event | 5 Years
  Time to re-hospitalization due to any cardiovascular event

OTHER OUTCOMES:
NT-pro-brain natriuretic peptide (NT-proBNP) levels | Baseline, discharge, 1, 3, and 6 month follow-up visits.
  NT-pro-brain natriuretic peptide (NT-proBNP) levels
Short Form 12 (SF-12) Questionnaire | Baseline (prior to the index STEMI), 1, 3, 6 and 12 month follow-up visits
  The SF-12 is a validated general quality of life self-administered instrument that has been used in various disease states.
Measurement of alginate in plasma and urine | Baseline, 5, 30 min, 1, 3, 8, 24, 48 hrs, 1, 3 month
  At selected sites, relatively intensive sampling: blood will be drawn just prior to deployment (0 hour), 5 and 30 minutes and 1, 3, 8, 24, 48 hrs post deployment or until discharge, whichever occurs first, and at 1 and 3 month follow-up visit.
  At selected sites, urine collection for measurements of alginate, 4 urine samples, will be collected at baseline (within 30 min prior to deployment), 0-8 hrs (from the time immediately following the device deployment through 8 hrs post deployment), 8 through 24 hours through post deployment, 24 through 48 hrs or discharge (whichever comes first). In addition, a urine sample will be taken at 1 and 3 month follow-up visits.
  Remaining sites: sparse sampling blood will be drawn at 1, 8 and 24 hours, 1 month and post-deployment.
Healthcare utilization | 6 and 12 month follow-up visits.
  The healthcare utilization and questionnaire consists of subject responses to questions regarding mobility, self-care, usual activities, pain, discomfort, anxiety and depression.
Anatomic endpoints | 4 to 6 hours following deployment, 1, 3 and 12 month follow-up visits
  Anatomic endpoints: ejection fraction, end systolic volume index, mitral regurgitation, diastolic function, sphericity index, wall thickness, wall motion score and left ventricular (LV) mass index derived from the echocardiogram.
Primary Safety Evaluation | 1 Year
  The following safety endpoints will be adjudicated by a Clinical Events Classification Committee:
  1. Death
  2. Recurrent myocardial infarction (MI) or target vessel revascularization or stent thrombosis
  3. Significant arrhythmia requiring therapy
  4. Myocardial rupture
Long-term Safety Evaluation | 1 year to 5 years after device deployment
  1. Death
  2. Need for devices for the management of congestive heart failure (CHF)
     * automated implantable cardiac defibrillator (AICD)
     * cardiac resynchronization therapy
     * left ventricular assist device (LVAD)
  3. Heart transplant
Continuous Electrocardiogram Cardiac Safety Endpoints | Baseline, prior to discharge, 1, 3 and 6 month follow-up visits
  * New ischemia by ST segment deviation
  * QT/QTcF (Fridericia's heart rate correction) before and 18 hours after procedure
  * Severe bradycardia or tachycardia, including sustained ventricular or supraventricular tachycardia, total beats in episodes of tachycardia, total pauses and newly paced beats.
Clinical Chemistry, Hematology, and Urinalysis panel | Clinical Chemistry, Hematology: Baseline, 8 hours (± 2 hours) post-deployment, 1, 3, and 6 month follow-up visits. Urinalysis : Baseline and discharge
  Chemistry panel - levels of albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen, calcium, serum chloride, bicarbonate, direct bilirubin, creatinine, γ-GT, glucose, lactate dehydrogenase, potassium, sodium, and total bilirubin.
  Hematology panel - hemoglobin, hematocrit, mean corpuscular volume (MCV), red blood cell count (RBC), white blood cell (WBC) levels (with 5 part differential), and platelet count.
  Urinalysis - pH, specific gravity, RBC, WBC, glucose, protein in the urine, and a Human chorionic gonadotropin (HCG) pregnancy test
Performance Goal and Study Success | Baseline to 6 months
  5 mL/m2 change or greater in LVEDVI in IK-5001 group vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (82):
- United States (16):
  - Cardiology, P.C., Birmingham, Alabama
  - Harbor - UCLA Medical Center, Torrance, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami Hospital, Miami, Florida
  - St. Vincent Medical Group Inc., Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore Medical Center Weiler Division, The Bronx, New York
  - East Carolina Heart Institute - ECHI, Greenville, North Carolina
  - Carl and Edyth Lindner Center for Research and Education @ Christ Hospital, Cincinnati, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
- Australia (7):
  - Princess Alexandra Hospital, Woolloongabba, Brisbane
  - Gold Coast Hospital, Southport, Queensland
  - The Queen Elisabeth Hospital, Woodville South, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - The Northern Hospital, Melbourne, Victoria
  - Flinders Medical Centre, Bedford Park
  - Royal Perth Hospital - Dept. of Cardiology, Perth
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - CHU du Sart Tilman, Liège
- Canada (7):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - York PCI Research, Newmarket, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Québec
  - Centre Hospitalier Universitaire de Sherbrooke, Québec
- France (9):
  - Hopital de Brive Service de Cardiologie, Brive-la-Gaillarde
  - Hopital Henri Mondor, Créteil
  - Hopital du Bocage Central, Dijon
  - CHU Grenoble - Hopital Michallon, Grenoble
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Nice Hopital Pasteur, Nice
  - Hopital Lariboisiere, Paris
  - Nouvel Hopital Civil, Strasbourg
  - CHU de Toulouse - Hopital Rangueil, Toulouse
- Germany (17):
  - Vivantes Netzwerk fur Gesundheit GmbH, Kinikum Neukolln, Berlin
  - Vivantes Humboldt-Klinikum, Berlin
  - Helios Klinikum Erfurt, Erfurt
  - Elisabeth-Krankenhaus, Essen
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Klinik fur Innere Medizin, Kardiologie, Jena
  - Klinik fur Kardiologie and Angiologie Universitatsklinikum, Kiel
  - University of Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Universitatsmedizin Mannheim, Mannheim
  - Klinikum der Universitat Munchen LMU, München
  - Stadtische Kliniken Neuss - Lukaskrankenhaus, Neuss
  - Klinikum Oldenburg gGmbH, Oldenburg
  - St. Marien-Krankenhaus Siegen gem. GMbH, Siegen
  - Krankenhaus Barmherzige Brüder Abt.Kardiologie und Pneumologie, Trier
  - Helios Klinikum Wuppertal, Wuppertal
- Israel (9):
  - The Edith Wolfson Medical Center, Holon, Tel Aviv
  - HaEmek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - B'nai Zion Medical Center, Haifa
  - Hadassah University Medical Center Jerusalem-Cardiology, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center - Tel Hashomer, Tel Litwinsky
- Poland (8):
  - UCK, Kliniczne Centrum Kardiologii, Gdansk
  - Centrum Interwencyjnego Leczenia Chorob Serca i Naczyn z Pododdzialem Kardiologii Interwencyjnej, Krakow
  - I Klinika Kardiologii i Elektrokardiologii lnterwencyjnej oraz Nadcisnienia Tetniczego CM UJ, Krakow
  - Oddzial Kardiologiczny Wojewodzki Specjalistyczny Szpital im. Bieganskiego w Lodzi, Lodz
  - Samodzileny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Samodzielny Publiczny Szpital Kliniczny nr 2 PUM w Szczecinie, Szczecin
  - Pracownia Kardiologii Inwazyjnej, Warsaw
  - Cetrainy Szpital Kliniczny MSWIA, Warsaw
- Spain (5):
  - Hospital del Mar/Passeig Maritim 25-29, Barcelona
  - Hospital Juan Ramon Jimenez, Huelva
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico de Santiago de Compostela, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei X, Chen S, Xie T, Chen H, Jin X, Yang J, Sahar S, Huang H, Zhu S, Liu N, Yu C, Zhu P, Wang W, Zhang W. An MMP-degradable and conductive hydrogel to stabilize HIF-1alpha for recovering cardiac functions. Theranostics. 2022 Jan 1;12(1):127-142. doi: 10.7150/thno.63481. eCollection 2022. PMID 34987638
- [Derived] Rao SV, Zeymer U, Douglas PS, Al-Khalidi H, White JA, Liu J, Levy H, Guetta V, Gibson CM, Tanguay JF, Vermeersch P, Roncalli J, Kasprzak JD, Henry TD, Frey N, Kracoff O, Traverse JH, Chew DP, Lopez-Sendon J, Heyrman R, Krucoff MW. Bioabsorbable Intracoronary Matrix for Prevention of Ventricular Remodeling After Myocardial Infarction. J Am Coll Cardiol. 2016 Aug 16;68(7):715-23. doi: 10.1016/j.jacc.2016.05.053. PMID 27515331
- [Derived] Frey N, Linke A, Suselbeck T, Muller-Ehmsen J, Vermeersch P, Schoors D, Rosenberg M, Bea F, Tuvia S, Leor J. Intracoronary delivery of injectable bioabsorbable scaffold (IK-5001) to treat left ventricular remodeling after ST-elevation myocardial infarction: a first-in-man study. Circ Cardiovasc Interv. 2014 Dec;7(6):806-12. doi: 10.1161/CIRCINTERVENTIONS.114.001478. Epub 2014 Oct 28. PMID 25351198